CLINICAL TRIAL: NCT03205501
Title: Molecular Fluorescence Endoscopy for the Detection of (Pre)Malignant Lesions in Barrett's Esophagus Using a Fluorescent Tracer 'EMI-137' Targeting c-Met: a Single-center Feasibility and Safety Study
Brief Title: Molecular Fluorescence Endoscopy of (Pre)Malignant Esophageal Lesions
Acronym: EAGLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL59628.042.16
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus; Esophageal Cancer; Dysplasia in Barrett Esophagus
Keywords: BE; EAC; HGD; Esophagus
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV-tracer EMI-137 (Experimental): * IV-administration of EMI-137: all patients will receive 0.13 mg/kg of the fluorescent tracer EMI-137 intravenously.
  * Molecular Fluorescence Endoscopy: approximately 2,5 hours after tracer administration, Molecular Fluorescence Endoscopy will be performed with additional measurements of fluorescence signals.
  Interventions: Drug: IV-administation of EMI-137; Device: Molecular Fluorescence Endoscopy platform

INTERVENTIONS:
Drug: IV-administation of EMI-137 — Intravenous administration of 0.13 mg/kg of the fluorescent tracer EMI-137 approximately 2.5 hours prior to the endoscopy procedure.
  Other Names: Tracer administation
Device: Molecular Fluorescence Endoscopy platform — A flexible fluorescence fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fiber-probe is inserted through the standard working-channel of the standard clinical endoscope. Fluorescence imaging will be performed prior to and post the endoscopic resection, during the same endoscopy procedure.
  Other Names: Fluorescence Endoscopy

SUMMARY:
To improve detection of esophageal (pre)malignant lesions during surveillance endoscopy of patients at risk of developing malignancies, for example in Barrett's Esophagus (BE), there is a need for better endoscopic visualization and the ability for targeted biopsies. Optical molecular imaging of neoplasia associated biomarkers could form a promising technique to accommodate this need. It is known that the biomarker c-Met is overexpressed in dysplastic and neoplastic areas in BE segments versus normal tissue and has proven to be a valid target for molecular imaging.

Edinburgh Molecular Imaging Ltd (EMI) has developed a fluorescent tracer specifically targeting c-Met by labeling a small peptide to a fluorescent fluorophore: 'EMI-137'. The investigators hypothesize that when EMI-137 is administered intravenously, it accumulates in c-Met expressing high grade dysplasia (HGD) and esophageal adenocarcinoma (EAC), enabling (early) cancer visualization using a newly developed fluorescent fiber-bundle. This hypothesis will be tested in the current pilot intervention study.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, eligible for a diagnostic and/or therapeutic endoscopy;
* At least a suspicion of low grade dysplasia (LGD) based on a prior endoscopy;
* World Health Organization (WHO) performance score of 0-2;
* Written informed consent;
* Mentally competent person that is able and willing to comply with study procedures;
* For female subjects who are of childbearing potential, are premenopausal with intact reproductive organs or are less than 2 years post-menopausal:

  * A negative serum pregnancy test prior to receiving the tracer;
  * Willing to ensure that she or her partner uses effective contraception during the trial and for 3 months thereafter.

Exclusion Criteria:

* Pregnancy or breast feeding;
* Advanced stage EAC patient not suitable for endoscopic resection;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent anticancer therapy (chemotherapy, radiotherapy, vaccines, immunotherapy) delivered within the last three months prior to the start of the treatment
* The subject has been included previously in this study or has been injected with another investigational medicinal product within the past six months.
* History of myocardial infarction (MI), Transient Ischemic Attack (TIA), CerebroVascular Accident (CVA), pulmonary embolism, uncontrolled congestive heart failure (CHF), significant liver disease, unstable angina within 6 months prior to enrollment.
* The subject had any significant change in their regular prescription or non-prescription medication between 14 days and 1 day prior to Investigational Medicinal Product (IMP) administration. Occasional use of analgesics, such as non-steroid anti-inflammatory drugs and/or paracetamol, was permitted at the discretion of the investigator. Use of hormonal contraceptives is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Tumor-to-background ratio that allows the in vivo detection of (pre)malignant lesions in patients with Barrett's Esophagus using molecular fluorescence endoscopy. | Day 1
  Calculation of the in vivo tumor-to-background ratio (> 1.5) based on fluorescence intensities in (pre)malignant lesions compared to surrounding healthy esophageal tissue.
Safety: the number of participants with symptoms or changes in vital signs (blood pressure, heart frequency and temperature) and/or (serious) adverse events that are related to administration of EMI-137. | Up to day 3

SECONDARY OUTCOMES:
The correlation of fluorescence signals to histopathology from (pre)malignant lesions and surrounding normal esophageal tissue. | Up to 1 year
Identification of fluorescence lesions and correlation with histopathology on subsequent biopsies in the resection surface after endoscopic mucosal resection. | Up to 1 year
Quantification of fluorescence signals in vivo and ex vivo of (pre)malignant lesions and normal esophageal tissue using multi-diameter single-fiber reflectance single-fiber fluorescence (MDSFR-SFF) spectroscopy. | Up to 1 year
Visualization of the localization and distribution patterns of EMI-137 in the esophagus using ex vivo fluorescence microscopy. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: W.B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen; G.M. van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No